CLINICAL TRIAL: NCT04832269
Title: Effects of a Multiple Sclerosis Relapse Therapy With Methylprednisolone (MP) During Pregnancy on Offspring Cognitive Function, Stress Sensitivity, Behaviour and Functional and Structural Brain Development
Brief Title: Effects of a Multiple Sclerosis Relapse Therapy on Offspring Neurocognitive Development and Behaviour
Acronym: MS-Children
Status: Recruiting | Type: Observational
Sponsor: Jena University Hospital (Other)
Collaborators: Ruhr University of Bochum (Other); Interdisciplinary Center of Clinical Research of the Medical Faculty Jena (Unknown); Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Principal Investigator, Florian Rakers, Principal Investigator, Jena University Hospital
Other Study IDs: ZKSJ0130
Record Dates: First submitted 2021-02-18; First posted 2021-04-05 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Multiple Sclerosis
Keywords: fetal programming; pregnancy; relapse therapy
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — GC receptor sensitivity, methylation of the GR-receptor gene
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MP exposed group: children and adolescents (aged 8 to 18 years) of mothers with prenatal exposition to MP in the context of an MS relapse therapy
  Interventions: Other: Exposure to methylprednisolone during pregnancy
- MP non-exposed group/control group: children and adolescents of mothers suffering from MS aged 8 to 18 years

INTERVENTIONS:
Other: Exposure to methylprednisolone during pregnancy — Exposure to methylprednisolone during pregnancy in the context of an MS relapse therapy
  Groups: MP exposed group

SUMMARY:
Introduction: Fetal exposure to glucocorticoids (GCs) used to induce fetal lung maturation in women threatened by premature labour is known to induce aberrations in brain development and stress sensitivity, cognitive dysfunction and neuro-psychiatric disorders in later life which all predict early brain ageing. Another common source of fetal GC exposure is the treatment of relapses in multiple sclerosis (MS), the most common neurological disease in young women. Despite the lack of studies, the 300-fold higher dosage of GCs for MS relapse treatment compared to obstetric indications is considered harmless for the fetus . Objectives: To examine the effects of GCs for MS relapse treatment during pregnancy on offspring structural and functional brain development, stress sensitivity, and cognitive and behavioural performance. Methods: Epidemiological multi-centre cohort study in 80 children and adolescents aged 8 to 18 years whose mothers received GCs to treat a MS relapse during pregnancy compared to unexposed participants. Expected Impact: Creating a guideline-changing evidence-based risk-benefit assessment regarding benefits of the MS relapse therapy for the mother and potential harm to the child.

DETAILED DESCRIPTION:
Introduction: Multiple Sclerosis (MS) affects 1 in 1,000 people in industrialised countries, mainly women of childbearing age. To prevent MS relapses, most patients receive disease-modifying therapies (DMTs). However, most DMTs - with the exception of interferons and glatiramer acetate - are not approved during pregnancy. Consequently, DMTs are regularly discontinued during pregnancy with a subsequently increased risk of relapses. Thus, relapses during pregnancy are a common phenomenon. The average relapse rate per year in pregnant MS patients not taking DMTs during the 1st and 2nd trimester is nearly identical to the pre-partum period after which it significantly declines during the 3rd Trimester. The German Neurologic Society estimates that approximately 25% of all pregnant women with MS will suffer a relapse during their pregnancy period(s).

It is generally recommended by European and US guidelines to treat MS relapses during pregnancy with the synthetic glucocorticoid (GC) methylprednisolone (MP), which is thought to be harmless for the unborn. However, regardless of the undoubtedly positive effects of GCs for MS relapse treatment, there is considerable doubt as to whether synthetic GCs are as low in side effects for the child as MS guidelines assume. The fetus develops in the presence of very low GC levels because it is unable to produce cortisol until the end of pregnancy and about 90% of maternal cortisol is being inactivated by the placental enzyme 11ß-HSD2. In contrast to maternal cortisol, synthetic GCs are no substrate for the placental enzyme 11ß-HSD2 and, thus, pass the placenta without being inactivated. Once within the fetal circulation, GCs interfere with the development of the fetal central nervous system (CNS). The effects of synthetic GCs on fetal development and health and disease in later life as well as the mechanisms mediating these effects are best characterised for betamethasone exposure to induce fetal lung maturation in babies threatening premature labour as this treatment is used in nearly 10% of all pregnancies. In various studies excess exposure to synthetic GCs is associated with reduced birth weight, altered fetal brain development e.g., by direct effect on neuro- and gliogenesis via anti-proliferative effects on neural stem/progenitor cells, and persisting functional changes of the stress axis with its two arms, the hypothalamus-pituitary-adrenal axis (HPAA) and the autonomic nervous system (ANS). Supraphysiological GC concentrations are also thought to reset the set point of the negative feedback regulation of the fetal HPAA which results in an increase of HPAA activity in later life. Increased HPAA activity has been associated with increased stress sensitivity and a number of behavioural changes and neuropsychiatric disorders including anxiety, depressive-like disorders, and attention deficit hyperactivity disorder (ADHD). The relationship between adverse environmental influences during critical periods of fetal life, such as exposure to excess GC, and offspring health in later life is the basis of the 'Fetal Programming' hypothesis.

A predecessor study of the investigators' work group tested the hypothesis that fetal betamethasone treatment impairs structural and functional brain development as well as stress sensitivity leading to disturbances in overall neurocognitive performance and behaviour in later life. It is noteworthy, that the dosage of betamethasone (2 x 12mg, 24h apart) was approximately 300-fold lower than the dosage used to treat MS relapses (1000mg over 3-5 days). As a major study outcome, the investigators noticed detrimental effects of prenatal betamethasone exposure on general cognitive ability at the age of 8 - 9 years. Intelligence quotient (IQ)-scores in children who were prenatally exposed to betamethasone were on average 10.5 points lower than in controls, with a large effect size of d = 0.68. Even though IQ-scores of betamethasone-exposed children were still within the expected population range, the investigators assume that this difference is clinically relevant and impedes future life success of the participants. In addition, children exposed to betamethasone showed a significant increase in ADHD related symptoms on the International Classification of Diseases (ICD)-10-based rating scale, the Diagnostik-System für psychische Störungen nach ICD-10 und DSM-5 für Kinder und Jugendliche-III, with a medium effect size of d = 0.51. Electroencephalographic (EEG) analysis showed that BM-exposed children had a higher spectral edge frequency at rest and during stress suggesting a reduced overall neuroelectric relaxation capacity. Heart Rate Variability (HRV) analysis revealed a resetting of the ANS in betamethasone-exposed children.

Objectives: The primary goal of this study is to examine the general cognitive ability as a marker of brain development of children of MS patients who received MP to treat an MS relapse during pregnancy. The secondary goals are to determine the effects of MP administered during pregnancy on offspring structural and functional brain development and neuropsychiatric and behavioural performance. Stress sensitivity and epigenetic changes of GC receptor function will be measured to determine underlying mechanisms.

The study is based on the following hypotheses:

Fetal exposure to MP during relapse treatment in pregnant MS patients leads to

* disturbances in structural and functional brain development due to the maturational potential of MP which induces asymmetries in the complex sequence of the maturation of cerebral functional systems with lifelong changes in brain function,
* permanent alterations in HPAA sensitivity and autonomic function which are associated with neuropsychiatric and behavioural disturbances in later life, and
* alterations in GC receptor function and methylation of the GC receptor gene (NR3C1) and the H19/IGF2 locus as the underlying mechanisms linking MP exposition during pregnancy and offspring cognitive and behavioural functioning in later life.

Methods: The investigators will carry out a multicentre, observational, cross-sectional study in children and adolescents aged 8 to 18 years. The study design is retrospective due to ethical considerations of withholding the standard relapse treatment and the long study duration of at least 10 years. Following recruitment, all participants will undergo the same examination procedures in one study visit consisting of two days. By extending the study visit to two days, the investigators ensure stress-free examinations. In general, day 1 and day 2 of the study visits take place in direct succession. However, in case of scheduling issues or if the children and their parents live close by and do not want to stay overnight, there may be a few days in between.

The sequence of examinations was chosen in such a way that blood sampling and neuropsychological examinations induce as little stress as possible for the participants.

1. Functional brain development: The investigators will apply state-of-the-art neurocognitive, behavioural and mental health measures to determine the stage of functional brain development: General cognitive ability (primary endpoint) is determined using German age-appropriate versions of the Reynolds Intellectual Assessment Scales and Screening (RIAS) intelligence test. Behaviour is measured using three external assessment questionnaires which are routinely used in clinics and the scientific community. The German rating scale Fremdbeurteilungsbogen für Aufmerksamkeitsdefizit-/Hyperaktivitätsstörungen (FBB-ADHS) is based on the ICD-10 criteria for ADHD and assesses inattentiveness, hyperactivity, and impulsivity. The child behaviour checklist (CBCL), an established diagnostic screening procedure, measures psychopathological abnormalities in children and adolescents. The strengths and difficulties questionnaire (SDQ) assesses children's strengths and weaknesses. The Continuous Performance Test (CPT) is a clinically and scientifically established instrument to detect selective attention, vigilance, and impulsive behaviour with sufficient reliability and validity. Motor development is assessed using the Movement Assessment Battery for Children - Second Edition (M-ABC 2), which allows a reliable and time-efficient assessment of motor-coordinative deficits.
2. Structural brain development: The stage of structural brain development will be quantified based on a volumetric T1-MRI standard sequence using markers such as gyrification and cortical thickness as well as the BrainAge Score, which was development by the investigators' research group. The investigators expect that prenatal MP has a significant effect on brain age since GCs accelerate tissue differentiation and maturation at the expense of tissue growth.
3. Stress sensitivity and autonomic function: The individual stress sensitivity including the function of the HPAA and the autonomic nervous system is examined using the Trier Social Stress Test (TSST). This is an established and commonly used tool for children to generate a reproducible psychophysiological stress response using a simulated examination situation. It comprises a 10 minute rest period and a task period consisting of five-minute story-telling and mental arithmetic periods, which is completed in front of an "examination committee". Saliva samples for measurement of cortisol levels and alpha-amylase are taken before and during the stress test to determine HPAA and sympathetic activity at rest and during activation. In addition, continuous electrocardiography (ECG) and EEG leads are performed. The autonomic activity is also determined using HRV analysis from the derived ECG based on established HRV standards as well as on innovative nonlinear information based approaches developed at the department. Autonomic activity reflected in HRV is a sensitive marker of disturbances in the neurodevelopmental trajectory. Neurophysiological activation is measured using power spectral and nonlinear EEG analysis techniques.
4. Mechanism: The investigators will determine GC receptor sensitivity and epigenetic changes of the NR3C1 promoter and the H19/IGF2 locus.

Expected Impact: The results of this study will improve the ability of clinicians to make an evidence-based benefit-risk assessment regarding the continuation of a DMT during pregnancy under consideration of its safety under 'real world' conditions in relation to the potential long-term risks of an acute relapse therapy with MP for the health of the unborn child in later life.

The investigators expect that the results will provide an additional argument (1) to continue immunomodulatory relapse prophylaxis, e.g. with interferons during pregnancy, especially in light of their recently recognized relative safety for the child, or (2) to choose a long-acting DMT such as cladribine that provides lasting protection from relapses during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* MS diagnosis was made based on the McDonald criteria valid at the time of diagnosis
* Written consent by the legal guardians of the participating child following a detailed oral and written education
* Exposed group (n=40): Children and adolescents (aged 8 to 18 years) of mothers with prenatal exposition to MP in the context of a MS relapse therapy
* Non-exposed group (n=40): Children and adolescents of mothers suffering from MS without MP therapy during pregnancy (aged 8 to 18 years) matched for age, gender and social background

Exclusion Criteria:

* Perinatal complications such as cerebral bleeding, neonatal intensive care with ventilation, prenatal therapy with glucocorticoids except for an MS relapse
* Maternal abuse of noxious agents during pregnancy
* Long-term glucocorticoid medication (e.g. asthma)
* Preterm births (before 36 weeks of pregnancy)
* Severe disease making an examination impossible (e.g. mental retardation)
* disease-modifying therapy during pregnancy

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population is composed of children aged 8 to 18 from mothers with multiple sclerosis who received methylprednisolone in pregnancy and children aged 8 to 18 from mothers with multiple sclerosis without methylprednisolone therapy during pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-10-19 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
General cognitive ability - Reynolds Intellectual Assessment Scales and Screening (RIAS) | approx. 30 - 40 min.
  Intelligence quotient as measured by RIAS, higher scores denote better outcome.

SECONDARY OUTCOMES:
Structural brain development - BrainAge score | approx. 20 min.
  Volumetric cranial MRI change in standard T1 sequences (Developmental biomarker)
Salivary cortisol decay curve | approx. 5 min. per swab
  Salivary cortisol concentration (nmol/l) before, during, and after Trier Social Stress Test
Salivary alpha-amylase | approx. 5 min. per swab
  Salivary alpha-amylase concentration (U/ml) before, during, and after Trier Social Stress Test
Heart rate variability | approx. 75 min.
  Heart rate variability (band power low frequency, high frequency, and ratio; msec^2/Hz) before, during, and after the Trier Social Stress Test
Spectral edge frequency in the EEG | approx. 75 min.
  Fast Fourier transformation to measure cerebral activity before, during, and after the Trier Social Stress Test
External assessment sheet for attention deficit / hyperactivity disorder (FBB-ADHS, German Version) | approx. 15 - 20 min.
  Questionnaire for parents assessing attention deficit hyperactivity disorder associated behaviour. Items based on symptoms of hyperkinetic disorder (International Classification of Diseases-10) and attention deficit hyperactivity disorder (Diagnostic and Statistical Manual of Mental Disorders-5). Higher scores denote worse outcome.
Child Behavior Checklist (CBCL/6-18R) | approx. 15 - 20 min.
  Questionnaire for parents assessing the child's behavioural symptoms on eight scales - (1) anxious/depressed, (2) withdrawn/depressed, (3) somatic complaints, (4) social problems, (5) thought, sleep, and repetitive behaviour problems, (6) attention problems, (7) rule-breaking behaviour, and (8) aggressive behaviour. Higher scores denote worse outcome.
Strengths and Difficulties Questionnaire (SDQ-Deu-S) | approx. 15 - 20 min.
  Brief screening questionnaire for parents assessing emotional and behavioural problems, hyperactivity and inattention, peer relationship problems, and prosocial behaviour. Higher score denote worse outcome.
Continuous Performance Test (CPT) | approx. 15 min.
  Computer-based test of selective attention, vigilance, and impulsivity, measured as reaction time, performance variability, and commission and omission errors. Higher scores denote poorer performance.
Emotional excitability scale from Personality questionnaire for children between 9 and 14 years (PFK 9-14, German Version) | approx. 15 min.
  Computer-based personality assessment reported by the child; for ages 9 - 14
Movement Assessment Battery for Children - Second Edition (M-ABC-2) | approx. 20 - 30 min.
  Motor impairment assessment for ages 3 - 16
Child anxiety test III (KAT-III, German version) | approx. 5 min. each
  State and trait anxiety in children aged 6 - 18 years; before and after the Trier Social Stress Test; higher scores denotes higher subjective anxiety

OTHER OUTCOMES:
Methylation of GR-receptor gene | approx. 10 min.
  DNA methylation at GC receptor gene NR3C1 and at the H19 locus

CONTACTS AND LOCATIONS:
Overall Officials: Florian Rakers, Principal Investigator — University Hospital Jena; Matthias Schwab, Prof. Dr., Study Director — University Hospital Jena
Locations (2):
- Germany (2):
  - Ruhr University of Bochum, Bochum
  - University Hospital Jena, Jena

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moisiadis VG, Matthews SG. Glucocorticoids and fetal programming part 1: Outcomes. Nat Rev Endocrinol. 2014 Jul;10(7):391-402. doi: 10.1038/nrendo.2014.73. Epub 2014 May 27. PMID 24863382
- [Background] Bloom SL, Sheffield JS, McIntire DD, Leveno KJ. Antenatal dexamethasone and decreased birth weight. Obstet Gynecol. 2001 Apr;97(4):485-90. doi: 10.1016/s0029-7844(00)01206-0. PMID 11275014
- [Background] Uno H, Eisele S, Sakai A, Shelton S, Baker E, DeJesus O, Holden J. Neurotoxicity of glucocorticoids in the primate brain. Horm Behav. 1994 Dec;28(4):336-48. doi: 10.1006/hbeh.1994.1030. PMID 7729802
- [Background] Antonow-Schlorke I, Helgert A, Gey C, Coksaygan T, Schubert H, Nathanielsz PW, Witte OW, Schwab M. Adverse effects of antenatal glucocorticoids on cerebral myelination in sheep. Obstet Gynecol. 2009 Jan;113(1):142-151. doi: 10.1097/AOG.0b013e3181924d3b. PMID 19104370
- [Background] van Dijk AE, van Eijsden M, Stronks K, Gemke RJ, Vrijkotte TG. Prenatal stress and balance of the child's cardiac autonomic nervous system at age 5-6 years. PLoS One. 2012;7(1):e30413. doi: 10.1371/journal.pone.0030413. Epub 2012 Jan 17. PMID 22272345
- [Background] Glover V, O'Connor TG, O'Donnell K. Prenatal stress and the programming of the HPA axis. Neurosci Biobehav Rev. 2010 Sep;35(1):17-22. doi: 10.1016/j.neubiorev.2009.11.008. Epub 2009 Nov 13. PMID 19914282
- [Background] Raikkonen K, Gissler M, Kajantie E. Associations Between Maternal Antenatal Corticosteroid Treatment and Mental and Behavioral Disorders in Children. JAMA. 2020 May 19;323(19):1924-1933. doi: 10.1001/jama.2020.3937. PMID 32427304
- [Background] Eriksson JG. The fetal origins hypothesis--10 years on. BMJ. 2005 May 14;330(7500):1096-7. doi: 10.1136/bmj.330.7500.1096. No abstract available. PMID 15891207
- [Background] Erhart M, Dopfner M, Ravens-Sieberer U; BELLA study group. Psychometric properties of two ADHD questionnaires: comparing the Conners' scale and the FBB-HKS in the general population of German children and adolescents--results of the BELLA study. Eur Child Adolesc Psychiatry. 2008 Dec;17 Suppl 1:106-15. doi: 10.1007/s00787-008-1012-1. PMID 19132310
- [Background] Schmeck K, Poustka F, Dopfner M, Pluck J, Berner W, Lehmkuhl G, Fegert JM, Lenz K, Huss M, Lehmkuhl U. Discriminant validity of the child behaviour checklist CBCL-4/18 in German samples. Eur Child Adolesc Psychiatry. 2001 Dec;10(4):240-7. doi: 10.1007/s007870170013. PMID 11794549
- [Background] Muris P, Meesters C, van den Berg F. The Strengths and Difficulties Questionnaire (SDQ)--further evidence for its reliability and validity in a community sample of Dutch children and adolescents. Eur Child Adolesc Psychiatry. 2003 Jan;12(1):1-8. doi: 10.1007/s00787-003-0298-2. PMID 12601558
- [Background] Schulz J, Henderson SE, Sugden DA, Barnett AL. Structural validity of the Movement ABC-2 test: factor structure comparisons across three age groups. Res Dev Disabil. 2011 Jul-Aug;32(4):1361-9. doi: 10.1016/j.ridd.2011.01.032. Epub 2011 Feb 16. PMID 21330102
- [Background] Franke K, Gaser C. Ten Years of BrainAGE as a Neuroimaging Biomarker of Brain Aging: What Insights Have We Gained? Front Neurol. 2019 Aug 14;10:789. doi: 10.3389/fneur.2019.00789. eCollection 2019. PMID 31474922
- [Background] Kirschbaum C, Pirke KM, Hellhammer DH. The 'Trier Social Stress Test'--a tool for investigating psychobiological stress responses in a laboratory setting. Neuropsychobiology. 1993;28(1-2):76-81. doi: 10.1159/000119004. PMID 8255414
- [Background] Schmidt K, Schwab M, Eiselt M, Kott M, Hoyer D, Zwiener U. Nonlinear modeling of different fetal and neo-natal behaviorial states. Pathophysiology. 1998;1001(5):257
- [Background] Frasch MG, Lobmaier SM, Stampalija T, Desplats P, Pallares ME, Pastor V, Brocco MA, Wu HT, Schulkin J, Herry CL, Seely AJE, Metz GAS, Louzoun Y, Antonelli MC. Non-invasive biomarkers of fetal brain development reflecting prenatal stress: An integrative multi-scale multi-species perspective on data collection and analysis. Neurosci Biobehav Rev. 2020 Oct;117:165-183. doi: 10.1016/j.neubiorev.2018.05.026. Epub 2018 May 30. PMID 29859198
- [Background] Kingwell E, Marriott JJ, Jette N, Pringsheim T, Makhani N, Morrow SA, Fisk JD, Evans C, Beland SG, Kulaga S, Dykeman J, Wolfson C, Koch MW, Marrie RA. Incidence and prevalence of multiple sclerosis in Europe: a systematic review. BMC Neurol. 2013 Sep 26;13:128. doi: 10.1186/1471-2377-13-128. PMID 24070256
- [Background] Confavreux C, Hutchinson M, Hours MM, Cortinovis-Tourniaire P, Moreau T. Rate of pregnancy-related relapse in multiple sclerosis. Pregnancy in Multiple Sclerosis Group. N Engl J Med. 1998 Jul 30;339(5):285-91. doi: 10.1056/NEJM199807303390501. PMID 9682040
- [Background] Society GN. Guidline for the treatment of Multiple Sklerosis. https://www.dgn.org/images/red_leitlinien/LL_2012/pdf/030-050l_S2e_Multiple_Sklerose_Diagnostik_Therapie_Archiv-min.pdf. Published 2012
- [Background] Dobson R, Dassan P, Roberts M, Giovannoni G, Nelson-Piercy C, Brex PA. UK consensus on pregnancy in multiple sclerosis: 'Association of British Neurologists' guidelines. Pract Neurol. 2019 Apr;19(2):106-114. doi: 10.1136/practneurol-2018-002060. Epub 2019 Jan 5. PMID 30612100
- [Background] Hagmann-von Arx P, Grob A. RIAS-Reynolds intellectual assessment scales and screening: deutschspra-chige Adaptation der Reynolds Intellectual Assessment Scales (RIAS) & des Reynolds Intellectual Screening Test (RIST) von Cecil R. Reynolds und Randy W. Kamphaus: Manual. Hans Huber; 2014
- [Background] Malik M. Heart rate variability: Standards of measurement, physiological interpretation, and clinical use: Task force of the European Society of Cardiology and the North American Society for Pacing and Electrophysi-ology. Annals of Noninvasive Electrocardiology. 1996;1(2):151-181
- [Derived] Kozik V, Schwab M, Thiel S, Hellwig K, Rakers F, Dreiling M. Protocol for a Cross-Sectional Study: Effects of a Multiple Sclerosis Relapse Therapy With Methylprednisolone on Offspring Neurocognitive Development and Behavior (MS-Children). Front Neurol. 2022 Apr 26;13:830057. doi: 10.3389/fneur.2022.830057. eCollection 2022. PMID 35557615
- See also: Official web page providing study information — http://www.ms-kinder.de